CLINICAL TRIAL: NCT03274973
Title: A Prospective Non-Interventional Study to Assess Long-term Effectiveness of Zomacton® and Factors Affecting Adherence in Patients With Growth Hormone Deficiency or Growth Retardation Due to Ullrich-Turner Syndrome
Brief Title: Study to Assess Long-term Effectiveness of Zomacton® and Treatment Adherence in Patients With Growth Hormone Deficiency or Ullrich-Turner Syndrome
Acronym: RAZANT
Status: Terminated | Type: Observational
Why Stopped: Insufficient, delayed recruitment of participants
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000302
Record Dates: First submitted 2017-08-29; First posted 2017-09-07 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Zomacton
  Interventions: Drug: Zomacton

INTERVENTIONS:
Drug: Zomacton — Injection

SUMMARY:
Assessment of long-term effectiveness of ZOMACTON in treatment of Growth Hormone Deficiency or growth retardation due to Ullrich-Turner Syndrome and assessment of compliance and adherence, optionally with the aid of an electronic app or patient diary.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (< 18 years) with growth hormone deficiency or growth retardation due to Ullrich-Turner-Syndrome
* Patients already receiving or who have been prescribed Zomacton® de novo according to its German label; the decision to prescribe Zomacton® was made independently from participation and prior to enrollment in this study.
* Patient and their parents (or legal representatives) who are willing and able to provide signed informed consent for use of their personal data.

Exclusion Criteria:

* Participation in an interventional clinical study within the last 30 days prior to baseline visit or during the follow-up period

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Linear growth (change in height) | Over the first 12 months (month 0, 3, 6, 9 and 12)
  Change in height defined as the change of the standard deviation score of body height vs. baseline

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Klinik fuer Allgemeine Paediatrie der Christian-Albrechts-Universitaet zu Kiel (there might be other sites in this country), Kiel, Germany